CLINICAL TRIAL: NCT04468802
Title: Do Childhood Measles and DTaP Vaccination Decrease the Mortality Rate Caused by SARS CoV-2 in OECD Countries?
Brief Title: Do Childhood Measles and DTaP Vaccination Decrease the Mortality Rate Caused by COVID-19 in OECD Countries?
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Guven, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSSEAH--0965
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Measles Vaccine; Mortality
MeSH Terms: conditions — COVID-19 | interventions — Mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Case fatality rate — Mortality rate caused by SARS CoV-2

SUMMARY:
Mortality rates caused by SARS CoV-2 differ between countries and this difference might be explained by several reasons. Childhood vaccination rate is thought to be one of them. Therefore present study aimed to examine the possible relationship between DTaP (diphtheria, tetanus, pertussis) and measles vaccination rates of Organization for Economic Co-operation and Development (OECD) countries and case fatality rate (CFR) caused by SARS CoV-2.

DETAILED DESCRIPTION:
The mortality rates caused by SARS CoV-2 differ between countries and this difference might be explained by several reasons. Childhood vaccination rate is thought to be one of them. Therefore present study aimed to examine the possible relationship between DTaP (diphtheria, tetanus, pertussis) and measles vaccination rates of Organization for Economic Co-operation and Development (OECD) countries and case fatality rate (CFR) caused by SARS CoV-2.A total of 32 OECD countries, of northern hemisphere, have been included in this study. Statistical analysis performed according to the CFR data of these countries based on SARS CoV-2. The CFR data calculated according to the total mortality count of a specific country for the 3-month period down from the date when first SARS CoV-2 case was observed.

ELIGIBILITY:
Inclusion Criteria:

* Children vaccinated in OECD countries in northern hemisphere

Exclusion Criteria:

* Non vaccinated children
* Southern hemisphere countries
* non-OECD countries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children vaccinated in OECD countries in northern hemisphere
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Case Fatality Rate | 4 months
  Mortality rate caused by SARS CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided